CLINICAL TRIAL: NCT00434915
Title: Does DHEA Enhance the Effects of Exercise in Postmenopausal Women?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-02; P01AG014383 (NIH)
Record Dates: First submitted 2007-02-12; First posted 2007-02-14 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Aging
MeSH Terms: interventions — Dehydroepiandrosterone

INTERVENTIONS:
Drug: DHEA

SUMMARY:
Dehydroepiandrostrone (DHEA) and its sulfated ester (DHEAS) are high circulating weak androgens which have been associated with conditions that accompany age-related decline such as sarcopenia, hyperinsulinemia, osteopenia, and cardiovascular disease. The decline in DHEA with age is particularly marked in postmenopausal women. Exercise has always been advocated in women; benefit has been demonstrated inmuscle, bone and lipid physiology, as well as perception of energy and sense of well-being. This study aims to explore the combined effect of both DHEA and exercise in postmenopausal women, age range 55-75 years old. Subjects will receive DHEA (50mg/day) or placebo for a 12-week period. At the beginning and conclusion of the study patients will undergo testing for muscle strength, body composition, VO2 max, insulin sensitivity, muscle biopsy with mitochondria enzyme measurements, and psychological analysis. Blood samples pre and post intervention will also be obtained and the level of selected anabolic markers, lipids, and androgenic and sex steroid levels will be assessed. For the twelve-week period, both placebo and DHEA treated participants will be involved in a resistance and aerobic exercise program coordinated through the GCRC and the Dan Abraham Healthy Living Center. Several correlations have been established with respect to exogenous DHEA administration in postmenopausal women. None have evaluated oral DHEA therapy in the setting resistance and aerobic exercise, key therapies advocated in postmenopausal women. As a plausible anabolic hormone DHEA is hypothesized to accentuate the effects of exercise as has been shown for testosterone. This study, as a randomized double-blind placebo controlled trial, will investigate the effects, if any, of a regimented exercise program and DHEA supplementation in postmenopausal women, specifically for evidence of enhancement of exercise effect by oral supplementation with DHEA in attenuating age-related decline

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be postmenopausal women between the ages of 60 and 75 years old.
* Women with levels of DHEA less than 110 mg will be selected.

Exclusion Criteria:

* Individuals with history or biochemical evidence of liver disease, cardiovascular disease (other than controlled hypertension); polycythemia, cerebrovascular disorders, or disorder of glucose metabolism with fasting hyperglycemia or hypoglycemia will be excluded.
* Use of psycotropic drugs within six months prior to enrollment
* History of severe depression or psychotic disorder
* Professional athletes or BMI greater than 30kg/m2
* Anyone who has been in a regular (greater than twice/weekly) exercise program for more than 2 months prior to the study
* Severe rheumatologic condition with chronic pain not well controlled.
* Use of DHEA, estrogen, progesterone, testosterone, corticosteroid products up to six months prior to study

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2003-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
physical performance (VO2 peak, muscle strength as measured by chest press, double knee extension, and isokinetic knee extension
quality of life
glucose and insulin metabolism
muscle protein synthesis
body composition

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States